CLINICAL TRIAL: NCT05088434
Title: Comparison of the Fecal Microbiota Transplantation and ACHIM Suspension for Manipulating the Gut Microbiota in Patients With Irritable Bowel Syndrome
Brief Title: Fecal Microbiota Transplantation and ACHIM for Manipulating Gut Microbiota in IBS Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016/1914
Record Dates: First submitted 2021-09-07; First posted 2021-10-22 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2021-08

CONDITIONS: Irritable Bowel Syndrome; Dysbiosis
Keywords: IBS; Fecal microbiota transplantation; ACHIM; Placebo; Gut microbiota
MeSH Terms: conditions — Irritable Bowel Syndrome; Dysbiosis

STUDY DESIGN:
Intervention Model Description: Double-blinded placebo-controlled study
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blinded placebo-controlled study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- donor FMT (Active Comparator): Fresh stool samples were obtained immediately from close family member (donor) before being re-transplanted into the patient through a gastroscope.
  Interventions: Dietary Supplement: Donor fecal microbiota transplantation
- ACHIM (Active Comparator): One vial of ACHIM suspension (ACHIM Biotherapeutics AB, Sweden), containing 30 x 109 colony forming unit (CFU) of bacteria, was given through the work channel of a gastroscope into the lower part of duodenum.
  Interventions: Dietary Supplement: Anaerobically Cultivated Human Intestinal Microbiota (ACHIM)
- Placebo (Placebo Comparator): Fresh stool samples were obtained from the patients themselves immediately before transplantation and re-transplanted through a gastroscope.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Anaerobically Cultivated Human Intestinal Microbiota (ACHIM) — One vial of ACHIM suspension (ACHIM Biotherapeutics AB, Vallingby, Sweden), containing 30 x 109 colony forming unit (CFU) of bacteria, was given through the work channel of a gastroscope into the lower part of duodenum.
  Arms: ACHIM
Dietary Supplement: Donor fecal microbiota transplantation — Only 60 ml of sterile 0.9% normal saline were added to a stool specimen, collected from the respective donor, with a weight of ~30 g and homogenized manually. Then 60 ml of feces-suspension (screened from the patients view) were instilled through the work channel of a gastroscope into the lower part of the duodenum.
  Arms: donor FMT
Dietary Supplement: Placebo — Only 60 ml of sterile 0.9% normal saline were added to the patient's own stool specimen with a weight of ~30 g and homogenized manually. Then 60 ml of feces-suspension (screened from the patients view) were instilled through the work channel of a gastroscope into the lower part of the duodenum.
  Arms: Placebo

SUMMARY:
The double-blinded placebo-controlled study compares the effect of fecal microbiota transplantation vs. Anaerobically Cultivated Human Intestinal Microbiota (ACHIM) or placebo (own feces) on manipulating the gut microbiota in patients with diarrhea-predominant irritable bowel syndrome (IBS).

DETAILED DESCRIPTION:
Fecal transplantation (FMT), the infusion of a fecal preparation from a healthy donor into the gastrointestinal tract of another human being is capable of altering the gut microbiome of the new host. There is speculation that human faeces from a healthy donor may constitute the ideal "probiotic", thus suggesting FMT as a treatment option for conditions where an altered microbiota has been detected, including irritable bowel syndrome (IBS) . Anaerobically Cultivated Human Intestinal Microbiota (ACHIM) is an alternative way to manipulate gut microbiota instead of FMT. ACHIM suspension is a natural ecosystem of normal intestinal bacteria cultivated and propagated regularly in the laboratory (in vitro). After 20 years of cultivation ACHIM has retained the same rich biodiversity as the original stool sample, originating from a healthy donor in 1995. ACHIM can restore the ecological balance of the gut when it has been disturbed (dysbiosis) e.g. after antibiotic treatment. ACHIM has until now been given to over 400 patients (most of them suffering from recurrent Clostridium difficile infection) without any serious side effects being observed. Microbiological tests have shown that ACHIM is a well-balanced functional microbiota, and contains the major bacterial phyla Firmicutes, Bacteroidetes, Proteobacteria and Actinobacteria .

Thus, in the present study aims at comparing these methods safety and efficacy in relieving symptoms in patients with IBS. Given the ethical concerns of unknown and long-term adverse effects of FMT therapy, only patients with moderate to severe symptoms will be included.

Aim:

The primary aim of this open pilot study was to compare these two gut manipulating methods (FMT and ACHIM) in IBS patients.

The secondary aims were as follows;

1. To evaluate and to compare the safety and efficacy of FMT and ACHIM suspension in relieving symptoms in patients with IBS.
2. To evaluate and to compare the FMT and ACHIM on quality of life.
3. To compare the detailed characterisation of microbial community composition (by means of 16S rRNA profiling) and determination of the kinetics of changes following FMT and ACHIM vs. placebo.

Study design Participants and sample size In a blind study, patients who meet the Rome III criteria for IBS with moderate to severe abdominal symptoms will be included. The patients will be randomised in three groups for receiving either FMT, ACHIM suspension or placebo (own feces), and they will be followed for 12 weeks with regard to efficacy and safety parameters, as well as analysis of faecal samples.

Donor screening:

Donors of fecal flora are healthy individuals living in the same household as the patients. All donors are screened before donation for previous exposure to contagious infectious agents. Screening of blood included serologic testing for hepatitis A, hepatitis B, hepatitis C, HIV, Epstein-Barr virus and cytomegalovirus. All donor stool samples are cultured for enteric bacterial pathogens and screened for viruses and parasites.

Study procedures Suspension of fresh feces from a close family member for FMT or ACHIM will be instilled into the duodenum via an endoscope. This route of administration has been safe in all studies.

* Faeces transplantation protocol: Fresh stool samples are obtained immediately before FMT. 60 ml of sterile 0.9% N-saline are added to a stool specimen with a weight of ~30 g and homogenized manually. Screened from the patients' view, 40 ml of faeces-suspension are instilled through the work channel of a gastroscope into the lower part of the duodenum, and thereafter flushed with 60 ml of sterile 0.9% N-saline.
* ACHIM transplantation protocol: The ACHIM suspension (ACHIM Biotherapeutics, Sweden) is given through the work channel of a gastroscope into the lower part of duodenum, and thereafter flushed with 60 ml of sterile 0.9% N-saline.
* Stool samples will be collected twice before study (week - 4 and -0-1), then after week 1, 4 and 12 and after 6 months. Donor feces for FMT will also be collected. Fresh frozen dry stool is sampled at all time points, aliquoted and stored at -80 degrees (<24 hours from production to delivery).
* Microbial DNA analyses: Microbiota analysis was performed using the Genetic Analysis (GA) map™ DysbiosisTest (Genetic Analysis AS, Oslo, Norway). The GA-test is based on regular molecular biology techniques, comprising fecal sample homogenization and mechanical bacterial cell disruption; combined with chemical cell lysis; automated total bacterial genomic DNA extraction using magnetic beads; 16S ribosomal ribonucleic acid (rRNA) polymerase chain reaction (PCR) DNA amplification covering the variable regions V3-V9; probe labelling by single nucleotide extension; hybridisation to complementary probes coupled to magnetic beads; and signal detection using BioCode 1000A 128-Plex Analyzer (Applied BioCode, Santa Fe Springs, California, USA). A Dysbiosis Index (DI) above 2 (maximum 5) indicate a microbiota that differs from the reference group (DI 1-2: non-dysbiosis, DI 3: moderate, DI 4-5: severe dysbiosis).
* Blood samples (Complete blood count, kidney and liver function tests) and urine analysis.
* Symptom and quality of life assessment: Gastrointestinal symptoms, bowel habits and quality of life will be recorded during a 12 week follow up period, at day 0, weeks 1, 4, 12 and 28 for symptom and quality of life assessment. The patients are asked to report the severity of global IBS symptoms and each of the symptoms (diarrhoea, bloating, flatulence and pain) during the preceding week, using a four-point scale (0 = none, 1 = mild, 2 = moderate, 3 = severe). IBS Symptom Severity Scale (IBS-SSS) contains 5 questions that are rated on a 100-point visual analogue scale (VAS) (the severity of abdominal pain, the frequency of abdominal pain, the severity of abdominal distension, dissatisfaction with bowel habits, and interference with quality of life). The score ranging is from 0 to 500, with a higher score indicating the worse condition (scores < 175 represent mild IBS symptoms, 175 - 300 represents moderate severity, > 300 represent severe IBS). A decrease of 50 points on the IBS-SSS has been shown to correlate with improvement in clinical symptoms.

Short form of Nepean Dyspepsia Index (SF-NDI) will be used to evaluate quality of life.

Statistical analyses:

Longitudinal analysis of microbiota composition will be performed with repeated measures ANOVA (for alpha diversity and bacterial abundances). If non-normal data, arcsine square root transformation or a nonparametric test will be used. Original donor and recipient stool microbiota will be compared (measures of alpha diversity and abundances of taxa) at baseline and at each recipient stool sampling time point using nonparametric or parametric methods.

Safety considerations:

Long experience has been gained during the past years at Haukeland University Hospital in performing FMT for treatment-resistant Cl. difficile enterocolitis and have developed an extensive program for identifying safe donors of faeces for FMT. Over the years, no serious side effects have occurred. The subset of IBS patients who are eligible for the study are typically patients with a heavy symptom burden, with few treatment alternatives. Therefore, the balance of safety concerns versus possibility of symptom improvement is considered to be positive, and will stress the importance of collecting safety data on FMT and ACHIM before this treatment is becoming more widely used.

ELIGIBILITY:
Inclusion criteria:

* Patients of age between 18-and 65 years.
* Have IBS-Symptom Severity Scale (IBS-SSS) score >175.
* All patients are required to have symptoms for at least 12 months, fulfilling the Rome III criteria with either diarrhoea-predominant irritable bowel syndrome (IBS-D) or mixed constipation and diarrhoea (IBS-M) with bloating or flatulence as predominant symptoms.
* All patients will undergo appropriate investigations to exclude organic disease.

Exclusion criteria:

* History of inflammatory bowel diseases, gastrointestinal malignancy, blood in stool
* Antibiotic use within 1 month prior to FMT
* Immunocompromised patient defined as taking immuno-suppressive medications
* History of opportunistic infections within 1 year prior to FMT, oral thrush, or disseminated lymphadenopathy.
* Patients who are scheduled for abdominal surgery.
* Pregnant or lactating women.
* Patients taking probiotics or taking antibiotics within 4 weeks prior to installation.

Inclusion criteria of donors for FMT:

* Close healthy, family members
* > 18 years old.

Exclusion criteria of donors for FMT:

* Pregnancy or lactation
* History of inflammatory bowel diseases, IBS, chronic abdominal pain, or gastrointestinal malignancy, diarrhea, blood in stool
* Antibiotic and pre/probiotic use within 1 month prior to FMT.
* Immunocompromised defined as taking immuno-suppressive medications
* History of opportunistic infections within 1 year prior to FMT, oral thrush, or disseminated lymphadenopathy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Gut microbiota analysis | 6 months
  Change in bacterial signals from baseline before transplantation with either donor-FMT, ACHIM of placebo to after transplantation at weeks 1, 4, 12 and 24, by using the GA-map Dysbiosis Test (Genetic Analysis AS, Oslo, Norway). The GA-test is based comprising fecal sample homogenization and mechanical bacterial cell disruption; combined with chemical cell lysis; automated total bacterial genomic DNA extraction using magnetic beads; 16S rRNA PCR DNA amplification covering the variable regions V3-V9; probe labelling by single nucleotide extension; hybridisation to complementary probes coupled to magnetic beads; and signal detection using BioCode 1000A 128-Plex Analyzer (Applied BioCode, Santa Fe Springs, California, USA). A Dysbiosis Index (DI) above 2 (maximum 5) indicated microbiota that differs from the reference group (DI 1-2: non-dysbiosis, DI 3: moderate, DI 4-5: severe dysbiosis).

SECONDARY OUTCOMES:
Irritable bowel syndrome Symptom Severity Scale (IBS-SSS) | 6 months
  Change in IBS-SSS scores at baseline before transplantation with either donor-FMT, ACHIM or placebo will be compared to after transplantation at weeks 1, 4, 12 and 24. IBS Symptom Severity Scale (IBS-SSS) contained 5 questions (the severity of abdominal pain, the frequency of abdominal pain, the severity of abdominal distension, dissatisfaction with bowel habits, and interference with quality of life) that were rated on a 100-point visual analogue scale (VAS). The scores ranging from 0 to 500, with a higher score indicating worse condition (scores < 175 represent mild IBS symptoms, 175 - 300 represents moderate severity, > 300 represent severe IBS). A decrease of 50 points on the IBS-SSS correlated with improvement in clinical symptoms.
Bristol stool form scale | 6 months
  Change in stool forms from baseline before transplantation with either donor-FMT, ACHIM or placebo will be compared to after transplantation at weeks 1, 4, 12 and 24. Bristol Stool Scale (BSS) classified human feces into seven consistency categories (1 for constipation and 7 for diarrhea).
Short form of Nepean Dyspepsia Index (SF-NDI) | 6 months
  Short form of Nepean Dyspepsia Index (SF-NDI) was used to evaluate quality of life in a 10-item questionnaire with 5 sub-scales each examining the influence of dyspepsia on domains of health in patients, namely tension/anxiety, interference with daily activities, disruption to regular eating/drinking, knowledge towards/control over disease symptoms and interference with work/study. Lower SF-NDI scores indicated increased quality of life .Changes in SF-NDI scores at baseline before transplantation with either donor-FMT, ACHIM or placebo will be compared to to after transplantation at weeks 1, 4, 12 and 24.
Eysenck Personality Questionnaire Neuroticism (EPQ-N-12_ | 6 months
  Eysenck Personality Questionnaire Neuroticism (EPQ-N-12) with a cut-off value of 4, scored neuroticism that is defined as a general tendency to emotional over reactivity or over responsiveness. Change in scores at baseline before transplantation with either donor-FMT, ACHIM or placebo will be compared to to after transplantation at weeks 1, 4, 12 and 24.
Hospital Anxiety and Depression Scale (HADS) | 6 months
  Hospital Anxiety and Depression Scale (HADS) where scores >8 in either subscale indicated anxiety or depression. Change in HAD scores at baseline before transplantation with either donor-FMT, ACHIM or placebo will be compared to after transplantation at weeks 1, 4, 12 and 24.

CONTACTS AND LOCATIONS:
Overall Officials: Trygve Hausken, M.D, Ph.D, Study Chair — Haukeland University Hospital; Tarek Mazzawi, M.D, Ph.D, Principal Investigator — Haukeland University Hospital
Locations (1):
- Haukeland Unversity Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No